CLINICAL TRIAL: NCT01511458
Title: Non-invasive Chromosomal Examination of Trisomy
Brief Title: Non-invasive Chromosomal Examination of Trisomy Study
Acronym: NEXT
Status: Completed | Type: Observational
Sponsor: Roche Sequencing Solutions (Industry)
Collaborators: Perinatal Quality Foundation: Nuchal Translucency Quality Review (Unknown)
Responsible Party: Sponsor
Other Study IDs: TD007
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Trisomy 21
Keywords: Pregnancy; Fetal aneuploidy; Trisomy 21; Down Syndrome; Prenatal screening; Non-invasive prenatal testing; First trimester; Combined screening; Nuchal translucency; PAPP-A; hCG; cell free DNA; cf DNA; DNA; Performance characteristics of non-invasive first trimester screening; Harmony Prenatal Test
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patient with a trisomy 21 pregnancy confirmed by genetic testing.
- Control: Patients without a trisomy 21 pregnancy confirmed by either genetic testing or a normal newborn phenotype.

SUMMARY:
The purpose of this blinded, multi-center, prospective, case-controlled study is to compare the Ariosa Harmony™ Prenatal Test for trisomy 21 detection with a standard first-trimester prenatal screening test consisting of serum screening (PAPP-A,free beta-hCG [β-hCG] or total hCG) and a nuchal translucency (NT) measurement (i.e. combined first trimester screening) in a general screened population.

The performance characteristics of these two test modalities will be assessed relative to the clinical reference standard of genetic analysis of the fetus or phenotypic characterization and genetic analysis of the newborn.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old and can provide informed consent.
2. Subject is planning a hospital delivery.
3. Subject has a singleton pregnancy with a documented gestational age between 10 weeks, 0 days, and 14 weeks, 2 days, inclusive, at the time of the study blood sample collection.
4. Subject is planning to undergo combined first trimester prenatal screening that includes NT measurement, and when indicated, serum screening with total or free β-hCG and PAPP-A.

Exclusion Criteria:

1. Subject has known aneuploidy.
2. Subject has active or history of malignancy requiring major surgery and/or systemic chemotherapy.
3. Subject has a twin demise at any gestational age. Twin demise includes any reductions, spontaneous or elective, after sonographic identification of a second (or more) gestational sac. Any clinical, sonographic, or other testing that suggests twin demise would serve as an exclusion criterion.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women presenting for combined first trimester screening as part of routine prenatal care
Sampling Method: Non-Probability Sample
Enrollment: 18955 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Difference in sensitivity and specificity of Ariosa Harmony™ Prenatal Test (AUCt) and combined first-trimester screening for detection of T21. | Enrollment to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Norton, MD, Principal Investigator — Stanford University; Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (36):
- United States (26):
  - Tucson Medical Center, Tucson, Arizona
  - East Bay Perinatal Associates, Oakland, California
  - Stanford University, Palo Alto, California
  - Perinatal Diagnostic Center, Riverside, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - The Institute of Prenatal Diagnosis and Reproductive Medicine, San Gabriel, California
  - Christiana Care Health System, Newark, Delaware
  - Altus Research, Lake Worth, Florida
  - Fetal Diagnostic Institute of the Pacific, Honolulu, Hawaii
  - Northshore University Health System, Evanston, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Brigham and Women's Hospital - Center for Fetal Medicine and Prenatal Genetics, Boston, Massachusetts
  - Minnesota Perinatal Associates, Minneapolis, Minnesota
  - Robert Wood Johnson School of Medicine, New Brunswick, New Jersey
  - St. Peters University Medical Center, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Northwest Perinatal Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson Univeristy Hospital, Philadelphia, Pennsylvania
  - Women's Health Care Group of Pennsylvania, Wynnewood, Pennsylvania
  - Partners in Obstetrics and Gynecology, Pawtucket, Rhode Island
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Hospitals Leuven, Leuven, Belgium
- Canada (4):
  - Early Risk Assessment Program - University of Alberta, Calgary, Alberta
  - Ottawa Hospital and Research Institute, Ottawa, Ontario
  - Mount Sinai University, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
- University of Perugia, Perugia, Italy
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
- Sweden (2):
  - Sahlgrenska University Medical Center, Gothenburg
  - Karolinska University Hospital, Stockholm

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. Guidelines for Perinatal Care, Sixth Edition, October 2007.
- [Background] Nicolaides KH. A model for a new pyramid of prenatal care based on the 11 to 13 weeks' assessment. Prenat Diagn. 2011 Jan;31(1):3-6. doi: 10.1002/pd.2685. No abstract available. PMID 21210474
- [Background] Malone FD, Canick JA, Ball RH, Nyberg DA, Comstock CH, Bukowski R, Berkowitz RL, Gross SJ, Dugoff L, Craigo SD, Timor-Tritsch IE, Carr SR, Wolfe HM, Dukes K, Bianchi DW, Rudnicka AR, Hackshaw AK, Lambert-Messerlian G, Wald NJ, D'Alton ME; First- and Second-Trimester Evaluation of Risk (FASTER) Research Consortium. First-trimester or second-trimester screening, or both, for Down's syndrome. N Engl J Med. 2005 Nov 10;353(19):2001-11. doi: 10.1056/NEJMoa043693. PMID 16282175
- [Background] Nicolaides KH, Spencer K, Avgidou K, Faiola S, Falcon O. Multicenter study of first-trimester screening for trisomy 21 in 75 821 pregnancies: results and estimation of the potential impact of individual risk-orientated two-stage first-trimester screening. Ultrasound Obstet Gynecol. 2005 Mar;25(3):221-6. doi: 10.1002/uog.1860. PMID 15736186
- [Background] Cicero S, Rembouskos G, Vandecruys H, Hogg M, Nicolaides KH. Likelihood ratio for trisomy 21 in fetuses with absent nasal bone at the 11-14-week scan. Ultrasound Obstet Gynecol. 2004 Mar;23(3):218-23. doi: 10.1002/uog.992. PMID 15027007
- [Background] Borrell A. The ductus venosus in early pregnancy and congenital anomalies. Prenat Diagn. 2004 Sep;24(9):688-92. doi: 10.1002/pd.958. PMID 15386454
- [Background] Faiola S, Tsoi E, Huggon IC, Allan LD, Nicolaides KH. Likelihood ratio for trisomy 21 in fetuses with tricuspid regurgitation at the 11 to 13 + 6-week scan. Ultrasound Obstet Gynecol. 2005 Jul;26(1):22-7. doi: 10.1002/uog.1922. PMID 15937972
- [Background] Sonek J, Borenstein M, Dagklis T, Persico N, Nicolaides KH. Frontomaxillary facial angle in fetuses with trisomy 21 at 11-13(6) weeks. Am J Obstet Gynecol. 2007 Mar;196(3):271.e1-4. doi: 10.1016/j.ajog.2006.10.891. PMID 17346551
- [Background] ACOG Committee on Practice Bulletins. ACOG Practice Bulletin No. 77: screening for fetal chromosomal abnormalities. Obstet Gynecol. 2007 Jan;109(1):217-27. doi: 10.1097/00006250-200701000-00054. PMID 17197615
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin No. 88, December 2007. Invasive prenatal testing for aneuploidy. Obstet Gynecol. 2007 Dec;110(6):1459-67. doi: 10.1097/01.AOG.0000291570.63450.44. PMID 18055749
- [Background] Ehrich M, Deciu C, Zwiefelhofer T, Tynan JA, Cagasan L, Tim R, Lu V, McCullough R, McCarthy E, Nygren AO, Dean J, Tang L, Hutchison D, Lu T, Wang H, Angkachatchai V, Oeth P, Cantor CR, Bombard A, van den Boom D. Noninvasive detection of fetal trisomy 21 by sequencing of DNA in maternal blood: a study in a clinical setting. Am J Obstet Gynecol. 2011 Mar;204(3):205.e1-11. doi: 10.1016/j.ajog.2010.12.060. Epub 2011 Feb 18. PMID 21310373
- [Background] Lo YM, Corbetta N, Chamberlain PF, Rai V, Sargent IL, Redman CW, Wainscoat JS. Presence of fetal DNA in maternal plasma and serum. Lancet. 1997 Aug 16;350(9076):485-7. doi: 10.1016/S0140-6736(97)02174-0. PMID 9274585
- [Background] Fan HC, Blumenfeld YJ, Chitkara U, Hudgins L, Quake SR. Noninvasive diagnosis of fetal aneuploidy by shotgun sequencing DNA from maternal blood. Proc Natl Acad Sci U S A. 2008 Oct 21;105(42):16266-71. doi: 10.1073/pnas.0808319105. Epub 2008 Oct 6. PMID 18838674
- [Background] Chiu RW, Chan KC, Gao Y, Lau VY, Zheng W, Leung TY, Foo CH, Xie B, Tsui NB, Lun FM, Zee BC, Lau TK, Cantor CR, Lo YM. Noninvasive prenatal diagnosis of fetal chromosomal aneuploidy by massively parallel genomic sequencing of DNA in maternal plasma. Proc Natl Acad Sci U S A. 2008 Dec 23;105(51):20458-63. doi: 10.1073/pnas.0810641105. Epub 2008 Dec 10. PMID 19073917
- [Background] Chiu RW, Sun H, Akolekar R, Clouser C, Lee C, McKernan K, Zhou D, Nicolaides KH, Lo YM. Maternal plasma DNA analysis with massively parallel sequencing by ligation for noninvasive prenatal diagnosis of trisomy 21. Clin Chem. 2010 Mar;56(3):459-63. doi: 10.1373/clinchem.2009.136507. Epub 2009 Dec 21. PMID 20026875
- [Background] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Background] Dhallan R, Guo X, Emche S, Damewood M, Bayliss P, Cronin M, Barry J, Betz J, Franz K, Gold K, Vallecillo B, Varney J. A non-invasive test for prenatal diagnosis based on fetal DNA present in maternal blood: a preliminary study. Lancet. 2007 Feb 10;369(9560):474-81. doi: 10.1016/S0140-6736(07)60115-9. PMID 17292767
- [Background] Tong YK, Jin S, Chiu RW, Ding C, Chan KC, Leung TY, Yu L, Lau TK, Lo YM. Noninvasive prenatal detection of trisomy 21 by an epigenetic-genetic chromosome-dosage approach. Clin Chem. 2010 Jan;56(1):90-8. doi: 10.1373/clinchem.2009.134114. Epub 2009 Oct 22. PMID 19850629
- [Background] Ghanta S, Mitchell ME, Ames M, Hidestrand M, Simpson P, Goetsch M, Thilly WG, Struble CA, Tomita-Mitchell A. Non-invasive prenatal detection of trisomy 21 using tandem single nucleotide polymorphisms. PLoS One. 2010 Oct 8;5(10):e13184. doi: 10.1371/journal.pone.0013184. PMID 20949031
- [Derived] Norton ME, Jacobsson B, Swamy GK, Laurent LC, Ranzini AC, Brar H, Tomlinson MW, Pereira L, Spitz JL, Hollemon D, Cuckle H, Musci TJ, Wapner RJ. Cell-free DNA analysis for noninvasive examination of trisomy. N Engl J Med. 2015 Apr 23;372(17):1589-97. doi: 10.1056/NEJMoa1407349. Epub 2015 Apr 1. PMID 25830321
- See also: Click here for more information about Ariosa Diagnostics — http://www.ariosadx.com
- See also: Click here to find more information about the Perinatal Quality Foundation — http://www.perinatalquality.com/